CLINICAL TRIAL: NCT03331822
Title: The Effects of Bright Light Exposure on ICU Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Rosengart, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRO17010109
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Circadian Rhythm Disorders; Sleep
Keywords: circadian; light therapy; ICU nurse
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: This is randomized crossover trial, in which each nursing subject will serve as his or her own control: i.e., matched. The subjects will be nurses from the 6FG Trauma Intensive Care Unit at UPMC Presbyterian hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light (Experimental): High illuminance ,white lights positioned at each nursing station throughout the hallway to generate a uniform exposure of approximately 1,000-3,000 lux.
  Interventions: Other: Bright Light
- No Light (No Intervention): Ambient, standard white fluorescent environmental light will serve as control.

INTERVENTIONS:
Other: Bright Light — high illuminance white lights positioned at each nursing station throughout the hallway to generate a uniform exposure of approximately 1,000-3,000 lux. To achieve this illuminance, a Day*Light Classic Light will be positioned at each nursing station in the ICU hallway.
  Arms: Light

SUMMARY:
In the majority of intensive care units, nurses work 12 hour shifts that consist of days and nights. Shift work outside of 6am-6pm has been reported to cause fatigue, induce sleep disorders, and cause metabolic disturbances. This shift to a nocturnal 'day' rather than diurnal, can result in reduced work performance, processing errors, accidents at work, absenteeism, and reduced quality of life. More chronically, those working at night have been shown to experience higher risks of heart disease, cancer and shorter median durations of life span. Much of this elevated risk is thought to be due to altered exposure to light, the dominant environmental cue regulating our circadian rhythms.

As diurnal organisms much of our biology is regulated by the solar day. Acutely, bright light exposure (i.e., sun) regulates the phase of the biological clock principally through the suppression of melatonin, which biologically mediates increased alertness and in essence, 'our daytime alertness'. During the night melatonin gradually increases and induces tiredness and ultimately sleep. This, in part, is biology behind the use of melatonin in those with sleep disturbances or to mitigate jet lag, with cross-continental or transoceanic flights.

In this study, the investigators will randomize nurses in the hospital to receive either high intensity white light (3,000 lux) or standard ambient white fluorescent (~400 lx) light for 10 hours during their night shift. This high illuminance light, rich in blue spectrum, is what diurnal creatures, like humans, are exposed to during the day. The lights may subsequently be equipped with blue filters (442 nm) to heighten the exposure to the rich blue spectrum light. Exposure will commence at the beginning of the night shift (~7pm) and continue for 10 hours. The rationale for terminating exposure prior to shift end is to foster an onset of sleep biology. At the end of each shift, the nurses will complete the Stanford Sleepiness Scale and the Psychomotor Vigilance Task (PVT). Saliva samples will be collected for melatonin level analysis and the nurses will complete sleep diaries at home. The investigators hypothesize that exposure to high intensity lighting during night shifts will reduce fatigue and enhance alertness and computational capacity that correlates with reduced melatonin.

DETAILED DESCRIPTION:
This is randomized crossover trial, in which each nursing subject will serve as his or her own control: i.e., matched. The subjects will be nurses from the 6FG Trauma Intensive Care Unit at UPMC Presbyterian hospital. The PI or co-investigator will approach each nurse prior to the initiation of this study to obtain informed consent. Each nurse subject works approximately 7-8 nights out of 18 shifts in each month. The duration of this study is 1 month.

Each subject will be exposed to either the intervention or control arm solely based upon nursing assignment. Currently, nurses are assigned to care for patient on either the F or G side of the 6FG ICU, and there will be no changes made to shift assignments. For the purposes of this study, the F wing of the ICU will be ambient, standard white fluorescent environmental light and serve as control. The G wing of the ICU will be equipped with high illuminance white lights positioned throughout the hallway to generate a uniform exposure of approximately 3,000 lux. The current evidence suggests that >2000 lux is needed to achieve biological effects. The lights used are identical to those commercially available for the treatment of seasonal affective disorder. There have been over 70 clinical trials and several meta-analyses that have demonstrated the efficacy of light therapy for SAD. Adverse events were not significantly different between the light therapy and control groups. Thus, nurses will be assigned to either intervention or control based upon their standard nursing assignments.

At the end of each shift, subjects will complete the Stanford Sleepiness Scale on paper. This is the gold standard for subjective sleepiness levels. It was developed by Hoddes et al (1973) and is a simple 7-point rating scale. The scale is well validated and has been used in over 100 clinical trials. In addition, they will next complete the Psychomotor Vigilance Task (PVT) on their computer in the ICU. This test is the standard objective measure of alertness and wakefulness. It has been employed as a marker of attention deficit in hundreds of studies to date. It is a 10 minute test in which the subjects look at a small rectangular screen and press the mouse every time a bright circle appears. The number of lapses (responses greater than 500 ms) is recorded. Subjects will be assessed a total of n=6 times during the period of study.

The quality of sleep the day following exposure to either intervention or control will be assessed through the use of a sleep diary. The Consensus Sleep Diary was developed in 2012 by a collaboration of insomnia experts. The subject will record what time they got into bed, time they went to sleep, how long to fall asleep, how many times they woke up, time they finally woke up, time they got out of bed, rate the quality of sleep, and how rested or refreshed they felt. Subjects will maintain 1 diary that will catalogue sleep during a total of n=6 night shifts.

The principle biologic mediator of sleep and wakefulness is melatonin. Saliva samples will be collected at the start of the shift (around 7pm) and at the end of the shift (around 7am). Samples will be stored at -80 degrees for future analysis. Nurses will be sampled a total of n=2 times. These samples will be stored for a maximum of 1 month. At the conclusion of the period of study and collection of all samples, which is estimated to be 1 month, all samples will be analyzed. No sample with be stored after analysis.

The subjects will complete the Stanford Sleepiness Scale on paper at the end of each shift. This is the gold standard for subjective sleepiness levels. It was developed by Hoddes et al (1973) and is a simple 7-point rating scale. The scale is well validated and has been used in over 100 clinical trials. In addition, they will next complete the Psychomotor Vigilance Task (PVT) on their computer in the ICU. This test is the standard objective measure of alertness and wakefulness. It has been employed as a marker of attention deficit in hundreds of studies to date. It is a 10 minute test in which the subjects look at a small rectangular screen and press the mouse every time a bright circle appears. The number of lapses (responses greater than 500 ms) is recorded.

The quality of sleep the day following exposure to either intervention or control will be assessed through the use of a sleep diary. The Consensus Sleep Diary was developed in 2012 by a collaboration of insomnia experts. The subject will record what time they got into bed, time they went to sleep, how long to fall asleep, how many times they woke up, time they finally woke up, time they got out of bed, rate the quality of sleep, and how rested or refreshed they felt.

The principle biologic mediator of sleep and wakefulness is melatonin. Saliva samples will be collected at the start of the shift (around 7pm), at 3am (normal melatonin peak time), and at the end of the shift (around 6am). Samples will be stored at -80 degrees for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* All ICU nurses working at the University of Pittsburgh Trauma ICU.

Exclusion Criteria:

* Not working nights

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task | Immediately at the end of the night shift worked.
  This test is the standard objective measure of alertness and wakefulness. It has been employed as a marker of attention deficit in hundreds of studies to date. It is a 10 minute test in which the subjects look at a small rectangular screen and press the mouse every time a bright circle appears. The number of lapses (responses greater than 500 ms) is recorded.
Stanford Sleepiness Scale | Immediately at the end of the night shift worked.
  It was developed by Hoddes et al (1973) and is a simple 7-point rating scale. The scale is well validated and has been used in over 100 clinical trials.

SECONDARY OUTCOMES:
Consensus Sleep Diary | Throughout the course of the study for the night immediately following the night shift worked.
  The Consensus Sleep Diary was developed in 2012 by a collaboration of insomnia experts. The subject will record what time they got into bed, time they went to sleep, how long to fall asleep, how many times they woke up, time they finally woke up, time they got out of bed, rate the quality of sleep, and how rested or refreshed they felt.
Salivary melatonin concentration | Immediately at teh end of the night shift worked.
  A saliva sample will be obtained immediately following the night shift worked. It will be assayed for melatonin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Matthew R. Rosengart, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griepentrog JE, Labiner HE, Gunn SR, Rosengart MR. Bright environmental light improves the sleepiness of nightshift ICU nurses. Crit Care. 2018 Nov 13;22(1):295. doi: 10.1186/s13054-018-2233-4. PMID 30424793